CLINICAL TRIAL: NCT04635501
Title: Prospective, Multicenter, Single Arm, Pre-CE Marked Study of the AbsorbaSeal (ABS 5.6.7) Vascular Closure Device
Brief Title: AbsorbaSeal (ABS 5.6.7) Vascular Closure Device Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ID3 Medical (Other)
Collaborators: CyndRx, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CP004CE
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ABS 5.6.7 (Experimental): Patients whose access site will be closed with the AbsorbaSeal 5.6.7 Vascular Closure Device
  Interventions: Device: ABS 5.6.7

INTERVENTIONS:
Device: ABS 5.6.7 — Patients whose access site will be closed with the ABS 5.6.7

SUMMARY:
This study investigates the efficacy and safety of the AbsorbaSeal (ABS 5.6.7.) Vascular Closure device (VCD) for the closure of access site of patients requiring percutaneous diagnostic or interventional procedures. An expected total of 50 patients will be enrolled in this study. A total of 12 patients (4 patients per site) will be treated as roll-in phase, prior to enrollment of the first patient. The primary objective of this study is to assess the safety and effectiveness of the ABS 5.6.7. VCD in sealing the femoral arterial access site following diagnostic or interventional peripheral or coronary procedures. Following physician training, patients will be enrolled. Efficacy and safety analyses will be based on these patients. Patients will be followed procedurally to discharge, at one month, (follow-up commitment). Secondary objectives are to further characterize adverse events (serious and non-serious), clinical utility measures and health-related quality of life.

DETAILED DESCRIPTION:
With the increased number of percutaneous interventions being performed in outpatient settings, there is a growing need to obtain safer, faster, and more secure hemostasis following these procedures. Due to its automatic deployment feature and simplicity in operation. AbsorbaSeal (ABS 5.6.7) will lead to more widespread use and improve patient outcomes. The active closure system used in the ABS 5.6.7 ensures a secure closure. The composition of the seal used is completely bio-absorbable and does not require the use of adjunct materials (i.e. collagen, sutures, staples, etc.) needed in many of the devices currently available.

Extensive laboratory testing, acute animal labs and deployment in chronic animal studies were performed with ABS 6. After a few device modification to create the improved ABS 5.6.7, only minimal confirmatory testing was performed with the current, modified ABS 5.6.7. The extensive test results on the previous device iterations are used to complete the confirmatory testing of the ABS 5.6.7 design.

The First in Man (FIM) trial (CP001) supports the initial safety and effectiveness of ABS 5.6.7 in humans (n=20) and was completed prior to application for a pivotal Investigational Device Exemption (IDE) Study in the United States and a CE Mark Study approval (CP004CE) in the European Union.

The primary objective of this study is to assess the safety and effectiveness of the ABS 5.6.7. Enrollment into this study will include anatomically eligible patients requiring diagnostic and interventional procedures. Patients will be followed procedurally to discharge, at one month, (follow-up commitment). Secondary objectives are to further characterize adverse events (serious and non-serious), clinical utility measures, and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, minimum age of 18
* Patient provides written Informed Consent
* Patient is scheduled for a peripheral diagnostic or interventional procedure
* Patient is able to undergo emergent vascular surgery if a complication related to the VCD necessitates such surgery
* Patient has a 6French arterial puncture located in the common femoral artery (CFA)
* Target vessel has a lumen diameter > 5 mm
* Patient is willing and able to comply with all Study visits and procedures and complete follow-up visit
* Catheterization procedure is planned and elective

Pre-Procedure Exclusion Criteria:

* Prior target artery closure with any closure device or closure with manual compression ≤ 30 days prior to the peripheral catheterization procedure
* History of significant bleeding or with any known or documented bleeding disorders, such as thrombocytopenia (with < 100,000 platelet count), von Willebrand disease, anemia (Hgb < 10 g/Dl, Hct < 30%), thrombasthenia, decreased fibrinogen (< 200 mg/Dl), and Factor V deficiency
* Acute ST-elevation myocardial infarction ≤ 48 hours prior to the peripheral catheterization procedure
* Ineligible for introducer sheath removal
* Thrombolytic therapy (e.g. streptokinase, urokinase, t-PA) ≤ 24 hours prior to the peripheral catheterization procedure
* Evidence of a preexisting hematoma, arteriovenous fistula, or pseudo-aneurysm at the access site prior to start of femoral artery closure procedure
* Prior femoral vascular surgery or vascular graft in region of access site or contralateral common femoral artery
* Targeted femoral artery is tortuous or requires a sheath length > 10 cm
* Pregnant or lactating
* Mean body mass index (BMI) > 35 kg/m²
* Existing nerve damage in ipsilateral limb
* Fibrotic, heavily calcified femoral artery within 10mm of the entry point
* Non-palpable pulses in affected access limb

Intra-Procedure Exclusion Criteria:

* Difficult insertion of procedural sheath, needle stick problems at the onset of the peripheral procedure or difficult insertion of ABS 5.6.7
* Procedural sheath placement either through superficial femoral artery or into the profunda femoris artery or placement at or distal to bifurcation of the superficial femoral artery and the profunda femoris artery
* Common femoral artery (CFA) puncture site located above the lowest sweep of the inferior epigastric artery; referred to as a "high stick"
* Common femoral artery (CFA) access puncture site located on the front wall that continues through the back wall of the targeted vessel; referred to as a "back wall stick"
* Common femoral artery (CFA) access puncture site with multiple punctures of the CFA in an attempt to gain access to the targeted vessel known as "multiple sticks"
* Common femoral artery (CFA) access puncture located in the side wall region of the targeted access vessel; referred to as a "side wall stick"
* Interventional procedures with multiple exchanges during the procedure that cause elongation and trauma to the vessel compromising the tight seal between the vessel and the sheath
* Hematoma developing during the course of the percutaneous procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Rate of major complications | Post-procedure follow up 30 ± 7 days
  Composite of (1) closure-related bleeding requiring transfusion, (2) closure related vascular injury requiring repair surgery, (3) new ipsilateral lower extremity ischemia causing a threat to viability of limb requiring surgical or endovascular intervention, (4) closure-related infection requiring intravenous antibiotics and/or extended hospitalization, (5) new onset closure-related neuropathy in the ipsilateral lower extremity requiring surgical repair, and (6) permanent closure-related nerve damage.
Time to hemostasis (TTH) after index procedure (min) | Intraoperative
  TTH is defined as elapsed time between ABS 5.6.7 removal and first observed hemostasis

SECONDARY OUTCOMES:
Rate of minor complications | Post-procedure follow up 30 ± 7 days
  Composite of (1) closure-related bleeding requiring > 30 min. of continual manual compression to achieve initial arterial hemostasis, (2) late closure-related arterial bleeding (following hospital discharge), (3) closure-related hematoma > 6 cm, (4) Ipsilateral lower extremity arterial emboli, (5) ipsilateral deep vein thrombosis, (6) closure-related vessel laceration, (7) access site wound dehiscence, (8) localized access site infection treated with intramuscular or oral antibiotics, (9) closure related arteriovenous fistula not requiring treatment, (10) closure related pseudo-aneurysm requiring thrombin injection or fibrin adhesive injection, (11) closure related pseudo-aneurysm not requiring treatment, and (12) new onset of transient access site closure related neuropathy in the ipsilateral lower extremity that is transient (> 24 hrs. and < 30 days) and does not require surgical repair
Device success | Within 5 minutes following ABS 5.6.7 deployment
  Device Success defined as the ability to deploy the implant and achieve arterial hemostasis with ABS 5.6.7 alone or with post hemostasis adjunctive manual compression for 5 minutes or less.
Procedure success | Post-procedure follow up 30 ± 7 days
  Procedure Success defined as attainment of final arterial hemostasis using any method.

CONTACTS AND LOCATIONS:
Overall Officials: Koen Deloose, MD, Principal Investigator — AZ Sint Blasius
Locations (2):
- Belgium (2):
  - O.L.V. Hospital, Aalst
  - A.Z. Sint-Blasius, Dendermonde